CLINICAL TRIAL: NCT03480334
Title: Abscopal Effect of Radiotherapy and Nivolumab in Relapsed Hodgkin Lymphoma After Anti-PD1 Therapy
Acronym: AERN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Paul Broeckelmann, Dr., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln 3140
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Nivolumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental): Nivolumab 240 mg i.v. at 2-weekly intervals combined with 20Gy radiotherapy (RT) to a preferably progressive and not pre-irradiated single lesion. Nivolumab will be continued for a maximum of 18 months or until disease progression or unacceptable toxicity.
  Interventions: Other: Nivolumab plus radiotherapy

INTERVENTIONS:
Other: Nivolumab plus radiotherapy — Nivolumab 240 mg i.v. at 2-weekly intervals combined with 20Gy radiotherapy (RT) to a preferably progressive and not pre-irradiated single lesion. Nivolumab will be continued for a maximum of 18 months or until disease progression or unacceptable toxicity.

SUMMARY:
The aim of the trial is to improve efficacy of nivolumab in patients with relapsed or refractory HL who recently progressed on anti-PD1 therapy. Nivolumab is highly effective and well tolerated in rrHL, nevertheless CR-rates are low and a considerable proportion of patients suffers from progressive disease. Localized RT induces an immunogenic effect which might work synergistically and facilitate augmented systemic (i.e. abscopal) responses in combination with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Progression of refractory or relapsed cHL during treatment with an anti-PD1 agent
* At least two distinct FDG-avid HL-lesions with at least 5 cm distance between them, and one of them considered eligible for irradiation with 20Gy based on localization and prior RT exposure
* Age at registration ≥ 18 years

Exclusion Criteria:

* Nodular-lymphocyte predominant HL (NLPHL) or composite/greyzone lymphoma
* Lymphoma involving the central nervous system
* Naïve to treatment with anti-PD1 targeting antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
Abscopal response rate (ARR-6) | 12 weeks
  Abscopal response rate (ARR-6) with abscopal response centrally confirmed as restaging result after RT to a single lesion and at least four but not more than six nivolumab infusions (RE-6 result)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne, I. Dept. of Medicine
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided